CLINICAL TRIAL: NCT01954147
Title: Umbilical Cord Mesenchymal Stem Cell Infusion With Liraglutide in Type 2 Diabetes Mellitus
Brief Title: Umbilical Cord Mesenchymal Stem Cells and Liraglutide in Diabetes Mellitus
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Diabetes Care Center of Nanjing Military Command (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: SC/GLP-1
Record Dates: First submitted 2013-08-13; First posted 2013-10-01 (Estimated); Last update posted 2014-02-20 (Estimated); Status verified 2014-02

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Glucagon-Like Peptide 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- SC-GLP-1 (Experimental): Umbilical Cord Mesenchymal Stem Cell Infusion Combined With Liraglutide
  Interventions: Drug: GLP-1; Biological: SC; Other: Standard Medical Treatment
- SC (Experimental): Umbilical Cord Mesenchymal Stem Cell Infusion
  Interventions: Biological: SC; Other: Standard Medical Treatment
- GLP-1 (Experimental): Liraglutide
  Interventions: Drug: GLP-1; Other: Standard Medical Treatment
- Control (Active Comparator): Standard Medical Treatment
  Interventions: Other: Standard Medical Treatment

INTERVENTIONS:
Drug: GLP-1 — GLP-1 therapy
  Arms: GLP-1; SC-GLP-1
Biological: SC — Stem cell infusion
  Arms: SC; SC-GLP-1
Other: Standard Medical Treatment — Standard Medical Treatment
  Other Names: SMT

SUMMARY:
Umbilical cord mesenchymal stem cells (SC) transplantation was a novel therapy for diabetes mellitus, with less side effects and more advantages. Clinical trials had verified that good metabolic control would be achieved when Liraglutide (GLP-1) was added to the conventional therapies. The investigators hypothesized that the combined therapy of umbilical cord mesenchymal stem cells transplantation and Liraglutide in type 2 diabetes mellitus will aid the differentiation of stem cells into insulin-producing cells, improve the survival of differentiated cells, protect the residual beta-cells and improve insulin secreting function, so as to achieve a favorable glucose homeostasis.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients age 35 to 65 years of age.
* Ability to provide written informed consent.
* Mentally stable and able to comply with the procedures of the study protocol.
* Clinical history compatible with type 2 diabetes (T2DM) as defined by ADA(1997) on the Diagnosis and classification of Diabetes Mellitus
* Basal C-peptide 0.5-2.0 ng/mL
* HbA1c ≥ 7.5 and ≤ 11% before standard medical therapy (SMT).
* Patients must have been treated with SMT for 1-4 months prior to matching. Insulin dose and metformin doses should be stable over 1 month prior to matching.
* HbA1c ≥ 7.5 and ≤ 10% at time of matching.
* Total insulin daily dose (TDD) at time of matching should not exceed 1.0 units/day/kg
* 18.5 kg/㎡≤BMI≤40.0kg/㎡

Exclusion Criteria:

* Abnormal liver function >2.5 x ULN
* Evidence of renal dysfunction:serum creatinine > 1.5 mg/dl (males) and 1.3 mg/dl (females).
* Gastrointestinal operation history.
* Type 1 Diabetes mellitus; DKA; secondary diabetes.
* Uncontrolled blood Pressure: SBP >180 mmHg or DBP >100 mmHg at the time of matching.
* Evidence of cardiovascular disease, existing congestive cardiac failure on physical exam and/or acute coronary syndrome in past 6 months.
* Presence of active proliferative diabetic retinopathy or macular edema.
* Any acute or chronic infectious condition that in the criteria of the investigator would be a risk for the patient.
* For female participants: Positive pregnancy test, presently breast-feeding, or unwillingness to use effective contraceptive measures for the duration of the study. For male participants: intent to procreate 3 months before or after the intervention or unwillingness to use effective measures of contraception. Oral contraceptives, Norplant?, Depo-Provera?, and barrier devices with spermicide are acceptable contraceptive methods; condoms used alone are not acceptable.
* Active infection including hepatitis C, HIV, or TB as determined by a positive skin test or clinical presentation, or under treatment for suspected TB.
* Subjects that are being treated with any medication that could interfere with the outcome of the study such as: Thiazolidinediones and other glucagon like peptide 1 (GLP-1) analogues (Exenatide, Byetta), Pramlintide (Amylin), Dipeptidyl-peptidase IV (DPP-IV) inhibitors (i.e. Sitagliptin, Januvia)
* Any known or suspected allergy to liraglutide or other relevant products.
* Evidence of thyroid adverse events (serum calcitonin increase, goiter, thyroid cancer, et al) or pancreatitis caused by other GLP-1 analogues.
* Subjects with past history or family history of Medullary Thyroid Carcinoma(MTC) or Multiple Endocrine Neoplasia Syndrome Type 2(MEN2) .

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
HbA1C | 1 year

SECONDARY OUTCOMES:
Fasting Blood Glucose | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Xiangjin Xu, Professor, Principal Investigator — Diabetes Care Center of Nanjing Millitary Command
Locations (1):
- Diabetes Care Center of Nanjing Military Command, Fuzhou, Fujian, China

REFERENCES:
- [Derived] Chen P, Huang Q, Xu XJ, Shao ZL, Huang LH, Yang XZ, Guo W, Li CM, Chen C. [The effect of liraglutide in combination with human umbilical cord mesenchymal stem cells treatment on glucose metabolism and beta cell function in type 2 diabetes mellitus]. Zhonghua Nei Ke Za Zhi. 2016 May 1;55(5):349-54. doi: 10.3760/cma.j.issn.0578-1426.2016.05.004. Chinese. PMID 27143183